CLINICAL TRIAL: NCT02857868
Title: A Phase I, Open-label, Multi-center, Single-dose Study to Evaluate the Pharmacokinetics of ABL001 in Healthy Subjects With Normal Hepatic Function and Subjects With Impaired Hepatic Function
Brief Title: A Trial to Evaluate the Pharmacokinetics of ABL001 in Healthy and Hepatic Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2103
Record Dates: First submitted 2016-04-27; First posted 2016-08-05 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2018-07

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; ABL001; Child-Pugh; healthy subjects with normal hepatic function
MeSH Terms: interventions — asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABL001 (Experimental)
  Interventions: Drug: ABL001

INTERVENTIONS:
Drug: ABL001

SUMMARY:
The main purpose of this study is to evaluate the effect of varying degrees of impaired hepatic function (by Child-Pugh classification) on the pharmacokinetics (PK) of ABL001 after a single oral dose.

ELIGIBILITY:
Key Inclusion criteria:

* Body mass index of 18-36 kg/m2, with body weight 50 kg and no more than 120 kg
* Vital signs (after at least 3 minutes rest in the supine position) within the following ranges (inclusive):

  * Oral body temperature between 35.0 °C - 37.5 °C (95.0-99.5°F)
  * Systolic BP ≥90 mmHg and ≤140 mmHg
  * Diastolic BP ≥60 mmHg and ≤90 mmHg for healthy subjects and 50-100 mmHg for subjects with impaired hepatic function (groups 2-4)
  * Pulse Rate: ≥50 and ≤90 bpm for healthy subjects (group 1) and ≥50 and ≤100 bpm for subjects with impaired hepatic function (groups 2-4)
* Healthy subjects with no clinically significant abnormalities as determined by past medical history, physical examination, vital signs, ECG, and clinical laboratory test
* Subjects with Child-Pugh Clinical Assessment Score as calculated per the Child-Pugh classification

Key Exclusion Criteria:

* Presence of clinically significant ECG abnormalities or a family history or presence of prolonged QT-interval syndrome
* History of cardiac disease
* Sexually active males must use a condom during intercourse while taking the drug and for 7 days after stopping
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs
* Administration of strong or moderate CYP3A4 inhibitors or inducers (including St John's wort) within 14 days prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Primary Pharmacokinetics (PK): Cmax | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Primary Pharmacokinetics (PK): AUClast | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Primary Pharmacokinetics (PK): AUCinf | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Secondary Pharmacokinetics (PK): Tmax | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Secondary Pharmacokinetics (PK): T 1/2 | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Secondary Pharmacokinetics (PK): CL/F | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects
Secondary Pharmacokinetics (PK): Vz/F | at pre- dose (0 hour), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours post-dose
  To evaluate the pharmacokinetics of a single oral dose of ABL001 in subjects with various degrees of impaired hepatic function (by Child-Pugh classification) relative to healthy subjects

SECONDARY OUTCOMES:
Percentage of plasma protein binding as expressed by unbound fraction in plasma | 2 hours post-dose
  To evaluate ABL001 plasma protein binding
ABL001 pharmacokinetic parameter - Cmax - based on unbound fraction in plasma | 2 hours post-dose
  Unbound fraction I plasma includes but is not limited to unbound Cmax (Cmax)
ABL001 pharmacokinetic parameter - AUClast - based on unbound fraction in plasma | 2 hours post-dose
  Unbound fraction I plasma includes but is not limited to unbound AUClast (AUClast)
ABL001 pharmacokinetic parameter - AUCinf - based on unbound fraction in plasma | 2 hours post-dose
  Unbound fraction I plasma includes but is not limited to unbound AUCinf (AUCinf)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - University of Miami / Clinical Research Services, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoch M, Sato M, Zack J, Quinlan M, Sengupta T, Allepuz A, Aimone P, Hourcade-Potelleret F. Pharmacokinetics of Asciminib in Individuals With Hepatic or Renal Impairment. J Clin Pharmacol. 2021 Nov;61(11):1454-1465. doi: 10.1002/jcph.1926. Epub 2021 Jul 16. PMID 34115385
- See also: Results for CABL001A2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17159